CLINICAL TRIAL: NCT04323358
Title: Agreement and Accuracy of Different Devices for Biometry Measurements in Patients With Cataract
Acronym: Comparison
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 1845/2019
Record Dates: First submitted 2020-03-17; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Cataract; Cornea; Surgery
MeSH Terms: conditions — Cataract; Corneal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Which eye as well as the order of devices and observer will be randomized. Randomization information will be put in a sealed envelope on screening date and opened right before measurements start.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IOL Master® 700 (Active Comparator): Biometry will be performed three times consecutively.
  Interventions: Diagnostic Test: Biometry; Diagnostic Test: Keratometry
- Pentacam® (Active Comparator): Keratometry will be performed three times consecutively.
  Interventions: Diagnostic Test: Keratometry
- Casia II® (Active Comparator): Keratometry will be performed three times consecutively.
  Interventions: Diagnostic Test: Keratometry
- Spectralis Anterion® (Active Comparator): Biometry will be performed three times consecutively.
  Interventions: Diagnostic Test: Biometry; Diagnostic Test: Keratometry

INTERVENTIONS:
Diagnostic Test: Biometry — Patients will be asked to place the chin in position and open their eyes wide. In between measurements, the patient will be arranged so his eyes are in one horizontal line and each time before measurement the patient will be asked to blink several times.
  Arms: IOL Master® 700; Spectralis Anterion®
Diagnostic Test: Keratometry — Patients will be asked to place the chin in position and open their eyes wide. In between measurements, the patient will be arranged so his eyes are in one horizontal line and each time before measurement the patient will be asked to blink several times.

SUMMARY:
The rationale of this study is to compare repeatability, reproducibility and agreement of three different AS-OCT devices and Pentacam.

The investigational devices are approved biometry and keratometry devices to perform biometric/keratometric measurements preoperatively before cataract surgery. The measurements are used to calculate the needed IOL power.

Measurements with all four devices will be performed 3 times consecutively by two trained observer. The order of the observer, the order of devices as well as the eye (left/right) is randomized.

Examinations will be implemented in accordance with the approved investigational plan on subjects and includes: repeated biometry/keratometry with four different devices

DETAILED DESCRIPTION:
The rationale of this study is to compare repeatability, reproducibility and agreement of both, AS-OCT(s) and Pentacam. In our department three different AS-OCT devices and a HR Scheimpflug imaging device are currently in use for clinical routine to measure the cornea. Among refractive and anterior segment surgeons, there is no preferred and accepted method for accurate measurements of the corneal curvature. The four diagnostic tools are based on different technical and physical imaging principles and to date only limited information on their comparability exist. One advantage of ASOCT represents faster imaging speed when compared to Scheimpflug imaging. Thus, imaging misalignment, segmentation errors and defocus aberration can most likely be avoided by AS-OCT. Chen et al demonstrated that HR Scheimpflug imaging measurements of CCT were systematically higher than the measurements provided by FD AS-OCT. Further, repeatability, reproducibility and agreement of AS-OCT and Scheimpflug imaging device will be assessed during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract
* Age 40 and older (females of childbearing age will be interviewed if pregnancy is possible)

Exclusion Criteria:

* Contact lens wear within 5 days
* Pathologic changes of the cornea, eye lid or conjunctiva on slit- lamp examination
* History of corneal ocular surgery
* Microphthalmus
* Recurrent intraocular inflammation of unknown etiology
* Blind fellow eye
* Uncontrolled systemic or ocular disease

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Agreement of the four devices measuring mean keratometry value. | 1 year
  The measured K-Value of each device and the k-values within one device will be compared

SECONDARY OUTCOMES:
Agreement of the four devices measuring mean steep keratometry value. | 1 year
  The measured steep K-Value of each device and the steep k-values within one device will be compared
Agreement of the four devices measuring mean flat keratometry value. | 1 year
  The measured flat K-Value of each device and the flat k-values within one device will be compared
Agreement of the four devices measuring mean true keratometry value. | 1 year
  The measured true K-Value of each device and the true k-values within one device will be compared
Agreement of the devices measuring mean axial length | 1 year
  The measured axial length of each device and the axial length within one device will be compared
Agreement of the devices measuring mean lens thickness | 1 year
  The measured lens thickness of each device and the measured lens thickness within one device will be compared
Agreement of the devices measuring mean white-to-white measurement | 1 year
  The measured white-to-white distance of each device and the measured white-to-white distance within one device will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Menapace, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna Allgemeines Krankenhaus, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No